CLINICAL TRIAL: NCT05812040
Title: Clinical Value of Breast High-Resolution MR Ductography in Patients With Pathological Nipple Discharge: A Prospective, Exploratory Diagnostic Study
Brief Title: Clinical Value of Breast High-Resolution MR Ductography in Patients With Pathological Nipple Discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yue Hu, Dr., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SYSKY-2023-122-02
Record Dates: First submitted 2023-03-20; First posted 2023-04-13 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Breast Neoplasms; Nipple Discharge
MeSH Terms: conditions — Breast Neoplasms; Galactorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRD + HR-MRD (Other)
  Interventions: Diagnostic Test: Magnetic Resonance Ductography (MRD); and High-Resolution Magnetic Resonance Ductography (HR-MRD)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Ductography (MRD); and High-Resolution Magnetic Resonance Ductography (HR-MRD) — all participants will receive Magnetic Resonance Ductography (MRD) and High-Resolution Magnetic Resonance Ductography (HR-MRD) examination, using breast dedicated coil and microscopic coil, respectively

SUMMARY:
Nipple discharge is one of the common symptoms of breast disease patients. Nipple discharge can be divided into physiological and pathological nipple discharge (PND). Among patients with PND symptoms who undergo biopsy, 5%-21% of them are malignant, and the risk of malignancy increases with age. The primary diagnostic imaging methods for PND patients include mammography and breast ultrasound. Nearly half of PND patients who undergo traditional mammography and ultrasound examination have negative findings, but this does not rule out the presence of malignant lesions. Central duct excision is the gold standard for PND diagnosis, but invasive surgery without imaging guidance can lead to some complications. Magnetic Resonance Ductography (MRD), which uses water imaging technology to visualize the inside of the duct without contrast injection, can show imaging features of ductal lesions such as filling defects, irregularities of duct walls, and ductal obstruction. However, previous studies have shown that the signal-to-noise ratio of MRD images needs to be improved. Microscopy coil has the characteristics of small voxels and high spatial resolution, making it suitable for high signal-to-noise ratio imaging of small superficial structures. This provides a hardware foundation for improving the quality of MRD images. Therefore, in this study, the investigators aim to use the 3T MR instrument and microscopy coil to perform non-invasive high-resolution Magnetic Resonance Ductography (HR-MRD) on PND patients to evaluate the ability of HR-MRD to detect PND causes and the imaging features of duct-related lesions on HR-MRD, to assist in the accurate diagnosis and treatment of PND.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 and 75 years old.
* Pathological nipple discharge patients who received treatment at Sun Yat-sen Memorial Hospital. The diagnostic criteria for pathological nipple discharge include unilateral, single duct orifice, and spontaneous discharge of serous or bloody fluid. Patients who meet any of the above criteria are considered as pathological discharge.
* Willing to sign an informed consent form for clinical research and undergo HR-MRD and MRD examination.

Exclusion Criteria:

* Patients who have undergone surgery on the nipple-areolar complex of the PND breast side within the past year.
* Patients who have claustrophobia or metal implants in their body, which are not suitable for MRI scans.
* Patients who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Analyze the sensitivity and specificity of HR-MRD in detecting lesions that require surgical excision in patients with PND | 15 months

SECONDARY OUTCOMES:
Analyze the PPV and NPV of HR-MRD in detecting lesions that require surgical excision in patients with PND | 15 months
The difference of detection sensitivity between HR-MRD and MRD in identifying lesions requiring surgical excision | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Yue Hu, MD., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seltzer MH, Perloff LJ, Kelley RI, Fitts WT Jr. The significance of age in patients with nipple discharge. Surg Gynecol Obstet. 1970 Sep;131(3):519-22. No abstract available. PMID 5454537
- [Background] Orel SG, Dougherty CS, Reynolds C, Czerniecki BJ, Siegelman ES, Schnall MD. MR imaging in patients with nipple discharge: initial experience. Radiology. 2000 Jul;216(1):248-54. doi: 10.1148/radiology.216.1.r00jn28248. PMID 10887256
- [Background] Kanemaki Y, Kurihara Y, Itoh D, Kamijo K, Nakajima Y, Fukuda M, Van Cauteren M. MR mammary ductography using a microscopy coil for assessment of intraductal lesions. AJR Am J Roentgenol. 2004 May;182(5):1340-2. doi: 10.2214/ajr.182.5.1821340. No abstract available. PMID 15100142
- [Background] Bhattarai N, Kanemaki Y, Kurihara Y, Nakajima Y, Fukuda M, Maeda I. Intraductal papilloma: features on MR ductography using a microscopic coil. AJR Am J Roentgenol. 2006 Jan;186(1):44-7. doi: 10.2214/AJR.04.1600. PMID 16357375
- [Background] Fu P, Kurihara Y, Kanemaki Y, Okamoto K, Nakajima Y, Fukuda M, Maeda I. High-resolution MRI in detecting subareolar breast abscess. AJR Am J Roentgenol. 2007 Jun;188(6):1568-72. doi: 10.2214/AJR.06.0099. PMID 17515378
- [Background] Hirose M, Nobusawa H, Gokan T. MR ductography: comparison with conventional ductography as a diagnostic method in patients with nipple discharge. Radiographics. 2007 Oct;27 Suppl 1:S183-96. doi: 10.1148/rg.27si075501. PMID 18180226
- [Background] Kanemaki Y, Kurihara Y, Okamoto K, Nakajima Y, Fukuda M, Maeda I, Akiyama F. Ductal carcinoma in situ: correlations between high-resolution magnetic resonance imaging and histopathology. Radiat Med. 2007 Jan;25(1):1-7. doi: 10.1007/s11604-006-0091-5. Epub 2007 Jan 25. PMID 17225046
- [Background] Zhu J, Kurihara Y, Kanemaki Y, Ogata H, Fukuda M, Nakajima Y, Maeda I. Diagnostic accuracy of high-resolution MRI using a microscopy coil for patients with presumed DCIS following mammography screening. J Magn Reson Imaging. 2007 Jan;25(1):96-103. doi: 10.1002/jmri.20809. PMID 17154376
- [Background] Bahl M, Baker JA, Greenup RA, Ghate SV. Evaluation of Pathologic Nipple Discharge: What is the Added Diagnostic Value of MRI? Ann Surg Oncol. 2015 Dec;22 Suppl 3:S435-41. doi: 10.1245/s10434-015-4792-9. Epub 2015 Aug 7. PMID 26249144
- [Background] Mann RM, Balleyguier C, Baltzer PA, Bick U, Colin C, Cornford E, Evans A, Fallenberg E, Forrai G, Fuchsjager MH, Gilbert FJ, Helbich TH, Heywang-Kobrunner SH, Camps-Herrero J, Kuhl CK, Martincich L, Pediconi F, Panizza P, Pina LJ, Pijnappel RM, Pinker-Domenig K, Skaane P, Sardanelli F; European Society of Breast Imaging (EUSOBI), with language review by Europa Donna-The European Breast Cancer Coalition. Breast MRI: EUSOBI recommendations for women's information. Eur Radiol. 2015 Dec;25(12):3669-78. doi: 10.1007/s00330-015-3807-z. Epub 2015 May 23. PMID 26002130
- [Background] Nicholson BT, Harvey JA, Patrie JT, Mugler JP 3rd. 3D-MR Ductography and Contrast-Enhanced MR Mammography in Patients with Suspicious Nipple Discharge; a Feasibility Study. Breast J. 2015 Jul-Aug;21(4):352-62. doi: 10.1111/tbj.12417. Epub 2015 Apr 16. PMID 25882883
- [Background] Berger N, Luparia A, Di Leo G, Carbonaro LA, Trimboli RM, Ambrogi F, Sardanelli F. Diagnostic Performance of MRI Versus Galactography in Women With Pathologic Nipple Discharge: A Systematic Review and Meta-Analysis. AJR Am J Roentgenol. 2017 Aug;209(2):465-471. doi: 10.2214/AJR.16.16682. Epub 2017 May 24. PMID 28537847
- [Background] Expert Panel on Breast Imaging:; Lee SJ, Trikha S, Moy L, Baron P, diFlorio RM, Green ED, Heller SL, Holbrook AI, Lewin AA, Lourenco AP, Niell BL, Slanetz PJ, Stuckey AR, Vincoff NS, Weinstein SP, Yepes MM, Newell MS. ACR Appropriateness Criteria(R) Evaluation of Nipple Discharge. J Am Coll Radiol. 2017 May;14(5S):S138-S153. doi: 10.1016/j.jacr.2017.01.030. PMID 28473070
- [Background] Gupta D, Mendelson EB, Karst I. Nipple Discharge: Current Clinical and Imaging Evaluation. AJR Am J Roentgenol. 2021 Feb;216(2):330-339. doi: 10.2214/AJR.19.22025. Epub 2020 Dec 9. PMID 33295815